CLINICAL TRIAL: NCT04543084
Title: Improving Home Program Practice for People With Language Disorders After Stroke
Brief Title: Home Program Practice for People With Language Disorders After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019/12/11
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Intervention Model Description: Single-subject Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Subject Design (Other): Each participant will go through a baseline phase and then an intervention phase.
  Interventions: Behavioral: Logbook

INTERVENTIONS:
Behavioral: Logbook — Participants will record practice in a logbook.

SUMMARY:
Logbooks are one of the most commonly used methods to both support and track adherence in research studies. This study will look at using logbooks to support adherence to reading practice for individuals with post-stroke aphasia. It is thought that using a logbook will increase practice time.

ELIGIBILITY:
Inclusion Criteria:

* at least 6 months post left hemisphere stroke with a diagnosis of aphasia
* must have self-reported interest in working to improve reading comprehension
* access to the Internet
* speak English as a primary language

Exclusion Criteria:

* significant visual or hearing impairment as determined by "aphasia-friendly" and age-appropriate screening
* actively receiving speech-language pathology services in which computerized or reading comprehension home practice activities are assigned/requested
* severe auditory comprehension impairment that limits understanding of one-step directions (i.e., Western Aphasia Battery-Revised sequential commands subtest score below 8).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Change in minutes of practice | Up to 11 weeks
  The number of minutes practiced
Change in percentage of adherence to practice goal | Up to 11 weeks
  The amount of practice compared to the goal

SECONDARY OUTCOMES:
Reading comprehension | At first session and at last session time in between up to 5 months
  As measured by performance on the Reading Comprehension Battery for Aphasia-2 (RCBA-2). A higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Elena V. Donoso Brown, PhD, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No